CLINICAL TRIAL: NCT06716229
Title: Relationship of Nutritional Support for Critically Ill Children With Clinical Outcomes in a Pediatric Hospital in Bolivia in 2025 (NutPeBol)
Brief Title: Relationship of Nutritional Support for Critically Ill Children With Clinical Outcomes in a Pediatric Hospital in Bolivia (NutPeBol)
Acronym: NutPeBol
Status: Not yet recruiting | Type: Observational
Sponsor: MPH D Raul Copana-Olmos (Other)
Collaborators: Universidad Mayor de San Simón (Other); Hospital del Nino Manuel Ascencio Villarroel (Other)
Responsible Party: Sponsor-Investigator, MPH D Raul Copana-Olmos, Assistant professor, Hospital del Nino Manuel Ascencio Villarroel
Organization: Hospital del Nino Manuel Ascencio Villarroel (Other)
Other Study IDs: 03FM24D008
Record Dates: First submitted 2024-10-30; First posted 2024-12-04 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: Critically Ill Children; Nutritional Support
Keywords: Critically Ill children; Nutritional support

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this observational study is to learn about the characteristics of nutritional support in critically ill children. The primary question to be answered is Is there an association between nutritional support of the critically ill child and clinical and hospital outcomes in children admitted to a pediatric referral center? Patients will be followed throughout their hospitalization, with a step-by-step evaluation of the nutritional support received through standard care and a review of the results obtained in the patients.

DETAILED DESCRIPTION:
The study aims to know the type and characteristics of nutritional support received by critically ill children hospitalized in Bolivian hospitals; to follow them during their hospitalization to verify their weight, nutritional status and the nutritional support they receive; to understand which types of nutritional support offer better clinical and hospital outcomes; finally, to be able to propose some guidelines to physicians, through guidelines or other tools for the dissemination of scientific information, in order to benefit more children.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to intensive care or intermediate care in hospital wards
* Complete clinical and anthropometric data.

Exclusion Criteria:

* Congenital or acquired chronic disease affecting growth (secondary malnutrition)
* On medication (corticosteroids, immunoglobulins, albumin)
* Burn patients, with prosthetic implants, postoperative of large tumor resections.
* Unknown history of pre-referral hospital management or hospitalized in other health facilities.

Ages: 1 Month to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Critically ill children with acute conditions who are admitted to the PICU, intermediate care or wards of a pediatric referral hospital
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-04-06 (Estimated); Primary Completion 2025-11-28 (Estimated); Study Completion 2025-12-19 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in mid-upper arm circumference (MUAC) <11.5 cm (115 mm), weight-for-height z-score (WHZ) <-3, or bilateral pitting edema in critically ill children admitted to a pediatric hospital. | From March 2025 to March 2026
  Participants who received nutritional support achieved changes from baseline in mid-upper arm circumference (MUAC) <11.5 cm (115 mm), weight-for-height z-score (WHZ) <-3, or bilateral pitting edema in critically ill children.

CONTACTS AND LOCATIONS:
Locations (2):
- Bolivia (2):
  - Hospital del Nino Manuel Ascencio Villarroel, Cochabamba, Cercado
  - Universidad Mayor de San Simon, Cochabamba, Cercado

IPD SHARING:
Plan to Share IPD: Yes
All underlying IPDs that result in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Starting in January 2026

REFERENCES:
- [Background] Amano K, Maeda I, Ishiki H, Miura T, Hatano Y, Tsukuura H, Taniyama T, Matsumoto Y, Matsuda Y, Kohara H, Morita T, Mori M; East-Asian collaborative cross-cultural Study to Elucidate the Dying process (EASED) Investigators. Effects of enteral nutrition and parenteral nutrition on survival in patients with advanced cancer cachexia: Analysis of a multicenter prospective cohort study. Clin Nutr. 2021 Mar;40(3):1168-1175. doi: 10.1016/j.clnu.2020.07.027. Epub 2020 Jul 31. PMID 32771283
- [Background] Mikhailov TA, Kuhn EM, Manzi J, Christensen M, Collins M, Brown AM, Dechert R, Scanlon MC, Wakeham MK, Goday PS. Early enteral nutrition is associated with lower mortality in critically ill children. JPEN J Parenter Enteral Nutr. 2014 May;38(4):459-66. doi: 10.1177/0148607113517903. Epub 2014 Jan 8. PMID 24403379
- [Background] Ward SL, Gildengorin V, Valentine SL, Sapru A, Curley MA, Thomas N, Willson DF, Flori HR. Impact of Weight Extremes on Clinical Outcomes in Pediatric Acute Respiratory Distress Syndrome. Crit Care Med. 2016 Nov;44(11):2052-2059. doi: 10.1097/CCM.0000000000001857. PMID 27355525
- [Background] Fraipont V, Preiser JC. Energy estimation and measurement in critically ill patients. JPEN J Parenter Enteral Nutr. 2013 Nov;37(6):705-13. doi: 10.1177/0148607113505868. Epub 2013 Oct 10. PMID 24113283
- [Background] Mtaweh H, Tuira L, Floh AA, Parshuram CS. Indirect Calorimetry: History, Technology, and Application. Front Pediatr. 2018 Sep 19;6:257. doi: 10.3389/fped.2018.00257. eCollection 2018. PMID 30283765
- [Background] Mehta NM, Bechard LJ, Cahill N, Wang M, Day A, Duggan CP, Heyland DK. Nutritional practices and their relationship to clinical outcomes in critically ill children--an international multicenter cohort study*. Crit Care Med. 2012 Jul;40(7):2204-11. doi: 10.1097/CCM.0b013e31824e18a8. PMID 22564954
- [Background] Chima L, Mulrooney HM, Warren J, Madden AM. A systematic review and quantitative analysis of resting energy expenditure prediction equations in healthy overweight and obese children and adolescents. J Hum Nutr Diet. 2020 Jun;33(3):373-385. doi: 10.1111/jhn.12735. Epub 2020 Feb 19. PMID 32073189
- [Background] Mehta NM, Skillman HE, Irving SY, Coss-Bu JA, Vermilyea S, Farrington EA, McKeever L, Hall AM, Goday PS, Braunschweig C. Guidelines for the Provision and Assessment of Nutrition Support Therapy in the Pediatric Critically Ill Patient: Society of Critical Care Medicine and American Society for Parenteral and Enteral Nutrition. JPEN J Parenter Enteral Nutr. 2017 Jul;41(5):706-742. doi: 10.1177/0148607117711387. Epub 2017 Jun 2. PMID 28686844
- [Background] Larsen BMK, Beggs MR, Leong AY, Kang SH, Persad R, Garcia Guerra G. Can energy intake alter clinical and hospital outcomes in PICU? Clin Nutr ESPEN. 2018 Apr;24:41-46. doi: 10.1016/j.clnesp.2018.02.002. Epub 2018 Mar 2. PMID 29576361
- [Background] Tume LN, Valla FV, Joosten K, Jotterand Chaparro C, Latten L, Marino LV, Macleod I, Moullet C, Pathan N, Rooze S, van Rosmalen J, Verbruggen SCAT. Nutritional support for children during critical illness: European Society of Pediatric and Neonatal Intensive Care (ESPNIC) metabolism, endocrine and nutrition section position statement and clinical recommendations. Intensive Care Med. 2020 Mar;46(3):411-425. doi: 10.1007/s00134-019-05922-5. Epub 2020 Feb 20. PMID 32077997
- [Background] Brossier DW, Tume LN, Briant AR, Jotterand Chaparro C, Moullet C, Rooze S, Verbruggen SCAT, Marino LV, Alsohime F, Beldjilali S, Chiusolo F, Costa L, Didier C, Ilia S, Joram NL, Kneyber MCJ, Kuhlwein E, Lopez J, Lopez-Herce J, Mayberry HF, Mehmeti F, Mierzewska-Schmidt M, Minambres Rodriguez M, Morice C, Pappachan JV, Porcheret F, Reis Boto L, Schlapbach LJ, Tekguc H, Tziouvas K, Parienti JJ, Goyer I, Valla FV; Metabolism Endocrinology and Nutrition section of the European Society of Pediatric and Neonatal Intensive Care (ESPNIC). ESPNIC clinical practice guidelines: intravenous maintenance fluid therapy in acute and critically ill children- a systematic review and meta-analysis. Intensive Care Med. 2022 Dec;48(12):1691-1708. doi: 10.1007/s00134-022-06882-z. Epub 2022 Oct 26. PMID 36289081
- [Background] Gold DL, Mihalov LK, Cohen DM. Evaluating the Pediatric Early Warning Score (PEWS) system for admitted patients in the pediatric emergency department. Acad Emerg Med. 2014 Nov;21(11):1249-56. doi: 10.1111/acem.12514. PMID 25377402